CLINICAL TRIAL: NCT02724449
Title: A Clinical Evaluation of 3M Cavilon Advanced Barrier Film for the Treatment of Incontinence Associated Dermatitis (IAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-348
Record Dates: First submitted 2015-05-28; First posted 2016-03-31 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Dermatitis
Keywords: IAD; Fecal incontinence
MeSH Terms: conditions — Dermatitis; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cavilon Advanced Barrier Film (Experimental): Cavilon Advanced Barrier Film applied to areas of IAD
  Interventions: Device: Cavilon Advanced Barrier Film

INTERVENTIONS:
Device: Cavilon Advanced Barrier Film — Cavilon Advanced Barrier Fim's application applied twice a week

SUMMARY:
The purpose of this study is to obtain information concerning the safety and effective use of a protective barrier film in patients experiencing severe incontinence associated dermatitis.

DETAILED DESCRIPTION:
This is an open label, non randomized prospective case series evaluating 3M Cavilon Advanced Barrier Film for the treatment of severe incontinence associated dermatitis (IAD) in the presence or absence of continued fecal or fecal and urinary incontinence. The product will be applied twice a week for a maximum duration of 3 weeks. Subjects will be followed twice a week until healing, for a maximum of 3 weeks or earlier, if discharged from the facility. During the study period, the frequency and intensity of their incontinence will be monitored, twice a week photographic documentation and IAD site assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject 18 years of age or older?
2. Is the subject in a facility providing nursing care 24h per day?
3. Does the subject have severe incontinence-associated dermatitis eg breached or denuded skin? The ideal candidate would have denudement present.
4. Is the subject willing to have photos taken of their skin exposed to incontinence and permit use of the photos in potential publications?
5. Is the subject willing to release rights to 3M for use of the photos?
6. Has the subject signed an Institutional Review Board-approved informed consent document and authorized the use and disclosure of protected health information? At NS-LIJ, only subjects who are capable of consenting are eligible to enroll. The study will not include participants with decisional impairment that would render them incapable of informed consent.

18 years or older

Exclusion Criteria:

Subjects are excluded from participation in this study if any of the answers to these questions is yes.

1. If female, is the subject pregnant or breast feeding or have they given birth within the 3 weeks preceding the screening visit?
2. Does the subject have a known allergy to acrylates or cyanoacrylate?
3. Does the subject have a current pressure ulcer in the area where the skin is affected by incontinence?
4. Does the subject have an active genital herpes infection?
5. Does the subject have a pre-existing abnormal skin disease on the treatment areas that may affect skin assessment?
6. Does the skin area involved in this study require treatment with a concomitant medication or product?
7. Has the subject been enrolled in any investigational study within 30 days of the Screening Visit?
8. Does the subject have any medical condition that in the opinion of the investigator should exclude him/her from participating in the study?
9. Has the subject received antifungal powders within 24 hours prior to enrollment?
10. Has the subject received cyanoacrylate based skin protectant to the affected areas (such as Marathon) within 72 hours prior to enrollment?
11. Is the facility unwilling to discontinue use for this subject of Dimethicone containing wipes on the area where the investigational device will be applied?
12. Is the facility unwilling to discontinue use for this subject of Chlorhexidine Gluconate wipes on the area where the investigational device will be applied?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gray M, Beeckman D, Bliss DZ, Fader M, Logan S, Junkin J, Selekof J, Doughty D, Kurz P. Incontinence-associated dermatitis: a comprehensive review and update. J Wound Ostomy Continence Nurs. 2012 Jan-Feb;39(1):61-74. doi: 10.1097/WON.0b013e31823fe246. PMID 22193141
- [Result] Doughty D, Junkin J, Kurz P, Selekof J, Gray M, Fader M, Bliss DZ, Beeckman D, Logan S. Incontinence-associated dermatitis: consensus statements, evidence-based guidelines for prevention and treatment, and current challenges. J Wound Ostomy Continence Nurs. 2012 May-Jun;39(3):303-15; quiz 316-7. doi: 10.1097/WON.0b013e3182549118. PMID 22572899
- [Result] Beeckman D, Schoonhoven L, Verhaeghe S, Heyneman A, Defloor T. Prevention and treatment of incontinence-associated dermatitis: literature review. J Adv Nurs. 2009 Jun;65(6):1141-54. doi: 10.1111/j.1365-2648.2009.04986.x. Epub 2009 Apr 3. PMID 19374674

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Study: No competitive products evaluated.
Period: Overall Study
Arm/Group | Open-label Study
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cavilon Advanced Barrier Film
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 70.9 [19 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Incontinence Associated Dermatitis Score
Description: Patients who were experiencing Incontinence Associated Dermatitis (IAD) from exposure to urine, stool or a combination of both urine & stool received an application of the barrier film every 72 hours. A skin assessment tool designed for IAD was used to document each patient's IAD score over time. The area scored was divided into 6 zones, l & r buttocks, L & right thighs, perianal & gluteal cleft. The % area within each zone with denudement was X by 9, redness was X by 3 and healthy skin X 1. The total score range of the 6 zones was 0-3654 with 3654 being worst case scenario.
  Improvement of IAD Score - At baseline (enrollment) the six zones were evaluated for % of denudement, redness, pink and healthy skin assessed. At the end of subject's participation, assessment were completed again to determine final score & change for improvement was measured by reduction in IAD score No improvement of IAD score - No change in score Progression of IAD score - Increase in IAD score
Time Frame: Baseline and end of treatment (up to 3 weeks)
Measure: Number; unit: participants
Arm/Group | Open Label Study
Number analyzed (Participants) | 16
participants
  Improved IAD score | 13
  No improvement of IAD score | 1
  Worsening of IAD score | 2

ADVERSE EVENTS:
Groups:
- Open-label Study: Single arm study
Arm/Group | Open-label Study
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Study (N=16)
MI (Cardiac disorders) | 1 (1) — One subject had an Myocardial infarction, not related to device.
full thickness wound (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No